CLINICAL TRIAL: NCT01824433
Title: A 8-week, Rater-blind, Active-controlled, Randomized Study to Compare the Effectiveness of Venlafaxine With Fluoxetine in the Treatment of Postmenopausal Women With Major Depressive Disorder
Brief Title: Comparison of Venlafaxine and Fluoxetine in the Treatment of Postmenopausal Women With Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, Head of Depression Center, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VFPWMDD
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Major Depression
Keywords: venlafaxine; fluoxetine; postmenopause; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Venlafaxine Hydrochloride; Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- venlafaxine (Active Comparator): venlafaxine 75-225mg qd
  Interventions: Drug: venlafaxine
- fluoxetine (Active Comparator): fluoxetine 20-60mg qd
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Drug: venlafaxine — venlafaxine 75-225mg qd
  Other Names: Efexor
  Arms: venlafaxine
Drug: fluoxetine — fluoxetine 20-60mg qd
  Other Names: Prozac
  Arms: fluoxetine

SUMMARY:
Women are more prone to depression at certain points of the life cycle, although the etiologic and therapeutic implications remain largely unknown1,2. It is reported that pre- and postmenopausal women have a significant difference in response to some antidepressants, within a large clinical trial data set3, 4. A growing number of researches indicate that a woman's hormonal status may influence response to different forms of antidepressant medication. Specifically, younger women appeared to respond better to monoamine oxidase inhibitors (MAOIs) and selective serotonin reuptake inhibitor (SSRIs), whereas men and older women have tended to have relatively better responses to tricyclic antidepressants (TCAs) 1-5. One difference between these classes of antidepressants is that the SSRIs are strongly serotoninergic, whereas TCAs have predominantly noradrenergic effects. One pooled analysis 6 suggests that older women (age ≥ 50) tend to respond poorer to SSRI, while this phenomenen was not observed with venlafaxine.

The antidepressive mechanism of venlafaxine that has both noradrenergic and serotonergic effects is superior to SSRIs. As a noradrenergic and serotonergic antidepressant, venlafaxinee has been demonstrated of significant advantages in response and remission rates compared with various SSRIs. As mentioned above, older women tend to have relatively better responses to TCAs which is predominantly noradrenergic antidepressant. Postmenopausal women with depression also would be predicted to respond better to an SSRI if administered along with hormone replacement therapy 6. This could be critical to understanding age difference in antidepressant responses across the life cycle because circulating estrogen levels may modulate central serotoninergic pathways. Therefore, it is presumed that antidepressants which enhance both serotonergic and noradrenergic neurotransmission, as venlafaxine, may be more effective than SSRIs for postmenopausal women with major depressive disorder.

DETAILED DESCRIPTION:
The study is designed as a multicenter, rater-blind, parallel-group, active-controlled, flexible dose, randomized trial in postmenopausal women who are recently experiencing major depressive disorder.

Patients will be female, aged 55 or older, outpatient or inpatient status, with diagnosis of major depressive episode (single or recurrent) by DSM-IV, the current depressive episode within 1 years. The patients should also have HAMD-24 total score≥20,a HAMD-24 Item 1 (depressed mood) score≥2 at screening and baseline.

The eligible subjects will be randomly assigned to 1 of 2 treatment groups with 1:1 allocation ratio: venlafaxine 75~225mg/d or fluoxetine 20~60mg/d. Treatment and observational duration will be 56 days (8 weeks).

Primary efficacy measure will be assessed based on the decrease of HAMD-24 from baseline to endpoint. The secondary efficacy measures are change from baseline to endpoint in CGI-S, CGI-I, and Pain VAS et al.

The safety in this study will be assessed by adverse event reporting, clinical laboratory measurements and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 50 or older, memopausal.
* Meet DSM-IV criteria for current unipolar major depressive disorder.
* The total score of the HAMD-24 is at least 20 at screening and baseline.
* The current depressive episode within 1 year.
* If recurrent depression, the remission of previous episode is at least 5 years from the current episode.
* Providing informed consent form to participate in the study by patients or their legal representatives.

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than major depressive disorder.
* Substance abuse or dependence.
* Patients were also excluded if they had any medical condition that would contraindicate the use of venlafaxine or fluoxetine.
* Organic mental disease, including mental retardation.
* History of clinically significant disease, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require treatment during the study.
* Use of psychiatric agents within 5 days prior to randomization.
* Have proved no response to venlafaxin or fluoxetine by previous treatment.
* Participation in another clinical study within 4 weeks (or longer time according to the local requirement)
* Has received ECT or MECT within 3 months prior to randomization.
* Significant risk of suicidal and/or self-harm behaviors.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Overall Improvement | from baseline to endpoint(Week 8)
  change of 24-item Hamilton Rating Scale for Depression total score

SECONDARY OUTCOMES:
Improvement of individual symptoms | from baseline to endpoint(week 8)
  the mean change of HAMD-24 subscale score in items 10, 11, 12, 13 (anxiety and somatizations) at endpoint

OTHER OUTCOMES:
Pain | from baseline to endpoint
  the mean change of Pain visual analog scale (Pain VAS）
safety outcome | From enrollment to endpoint (Week 8)
  the proportion of patients who discontinue due to lack of efficacy or intolerability

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D.,Ph.D, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou J, Wang X, Feng L, Xiao L, Yang R, Zhu X, Shi H, Hu Y, Chen R, Boyce P, Wang G. Venlafaxine vs. fluoxetine in postmenopausal women with major depressive disorder: an 8-week, randomized, single-blind, active-controlled study. BMC Psychiatry. 2021 May 19;21(1):260. doi: 10.1186/s12888-021-03253-8. PMID 34011310